CLINICAL TRIAL: NCT01786551
Title: Effect of Eplerenone on Postprandial Inflammatory Response in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gail Kurr Adler, Associate Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010P002191
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Systemic Proinflammatory State
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eplerenone (Experimental): Eplerenone 50 mg daily for 14 days
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — 50 mg daily for 14 days

SUMMARY:
The purpose of this study is to investigate the effect of mineralocorticoid receptor (MR) blockade in healthy participants in a systemic proinflammatory state after a meal high in fat and glucose, which is associated with the pathogenesis of atherosclerosis.

Participants will include normal-weight, healthy males (Body Mass Index (BMI) ≤ 25 kg/m^2) between the ages of 18-45, without hypertension and clinical evidence of metabolic, cardiovascular or any other kind of diseases. After a 12-hour (h) fast, participants will be assigned to a combination of oral fat-loading test (OFLT) and oral glucose tolerance test (OGTT) (day 1), followed by a two-week treatment with 50 mg eplerenone. After two weeks, participants will receive the second OFLT/OGTT treatment (day 15). Starting 5 days prior to the first intervention (day1), the participant's usual diet (ad lib) will be supplemented with 2 bullion broths each day. Standardization of sodium intake is necessary as variations in dietary sodium intake may affect outcome measures. We will evaluate the following parameters at day 1 and day 15 of the study. Prior to OFLT/OGTT, and 2h, 4h thereafter, we will measure a parameter of vascular and systemic inflammation: interleukin-6 (IL-6).

ELIGIBILITY:
Inclusion Criteria:

* male
* 18-45 years
* BMI between 20-25 kg/m^2

Exclusion Criteria:

* evidence of cardiovascular, hepatic, renal [estimated glomerular filtration rate (GFR) <60 millimeter/minute (ml/min)] or any other organ system disease
* Blood pressure equal to or less than 90/60 mmHg
* prescription or herbal medications
* smoking
* alcohol consumption of more than 2 drinks per day
* dietary supplements

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail K Adler, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Krug AW, Stelzner L, Rao AD, Lichtman AH, Williams GH, Adler GK. Effect of low dose mineralocorticoid receptor antagonist eplerenone on glucose and lipid metabolism in healthy adult males. Metabolism. 2013 Mar;62(3):386-91. doi: 10.1016/j.metabol.2012.08.011. Epub 2012 Sep 21. PMID 23006216

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eplerenone
Started | 16
Completed | 14
Not Completed | 2
Not completed — Participant withdrew consent | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who completed the study and had glucose data available.
Arm/Group | Eplerenone
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Vascular and Systemic Inflammation as Measured by Interleukin-6 (IL-6) Serum Levels
Description: At Visit 1, blood was drawn before and then 2h and 4h after a high-fat/high-glucose meal (50 g fat, 75 g glucose). Participants then followed a low-dose eplerenone treatment (50 mg daily) for 14 days. At Visit 2, blood was drawn again before, 2h, and 4h after a high-fat/high-glucose meal after 14 days.
Time Frame: Baseline, 2 hours, and 4 hours, measured before and after 2 weeks of eplerenone treatment
Population: Data reported for evaluable participants only. All participants who completed the study and had glucose data available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eplerenone
Number analyzed (Participants) | 13
ng/mL
  Pre-eplerenone, baseline: number analyzed (Participants) | 11
  Pre-eplerenone, baseline | 1.70 (0.93)
  Pre-eplerenone, 2 hours: number analyzed (Participants) | 10
  Pre-eplerenone, 2 hours | 1.51 (0.73)
  Pre-eplerenone, 4 hours: number analyzed (Participants) | 12
  Pre-eplerenone, 4 hours | 1.65 (0.79)
  Post-eplerenone, baseline: number analyzed (Participants) | 11
  Post-eplerenone, baseline | 1.78 (0.85)
  Post-eplerenone, 2 hours: number analyzed (Participants) | 9
  Post-eplerenone, 2 hours | 1.47 (0.93)
  Post-eplerenone, 4 hours: number analyzed (Participants) | 12
  Post-eplerenone, 4 hours | 1.75 (0.96)

2. Secondary Outcome: Post-prandial Glucose Serum Levels
Description: as for outcome 1
Time Frame: Baseline, 2 hours, and 4 hours, measured before and after 2 weeks of eplerenone treatment
Population: Data reported for evaluable participants only. All participants who completed the study and had glucose data available.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Eplerenone
Number analyzed (Participants) | 13
mg/dl
  Pre-eplerenone, baseline | 91 (7)
  Pre-eplerenone, 2 hours | 105 (28)
  Pre-eplerenone, 4 hours | 93 (17)
  Post-eplerenone, baseline | 89 (12)
  Post-eplerenone, 2 hours | 102 (21)
  Post-eplerenone, 4 hours | 92 (20)

3. Secondary Outcome: Post-prandial Insulin Serum Levels
Description: as for outcome 1
Time Frame: Baseline, 2 hours, and 4 hours, measured before and after 2 weeks of eplerenone treatment
Population: Data reported for evaluable participants only. All participants who completed the study and had glucose data available.
Measure: Mean (Standard Deviation); unit: uU/ml
Arm/Group | Eplerenone
Number analyzed (Participants) | 13
uU/ml
  Pre-eplerenone, baseline | 4.5 (3.6)
  Pre-eplerenone, 2 hours | 33.0 (45.7)
  Pre-eplerenone, 4 hours | 10.4 (10.7)
  Post-eplerenone, baseline | 5.7 (8.7)
  Post-eplerenone, 2 hours: number analyzed (Participants) | 11
  Post-eplerenone, 2 hours | 23.2 (21.5)
  Post-eplerenone, 4 hours: number analyzed (Participants) | 12
  Post-eplerenone, 4 hours | 8.7 (6.2)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: An adverse event (AE) is any untoward or unfavorable medical occurrence in a human subject including any abnormal sign, symptom or disease, whether or not associated with the subject's participation in the research. Unexpected and related/possibly research-related AEs were to be reported to the institutional review board (IRB). Expected AEs (documented in the protocol), were not reported to the IRB.
Arm/Group | Eplerenone
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No